CLINICAL TRIAL: NCT02591914
Title: An Open-Label Investigator Sponsored Trial to Investigate the Safety, Tolerability and Development of Subfoveal Fibrosis By Intravitreal Administration of Altering Regimens of Fovista and Anti-VEGF Therapy in Subjects With Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Retinal Consultants of Arizona (Other)
Collaborators: Ophthotech Corporation (Industry)
Responsible Party: Principal Investigator, Pravin Dugel, MD, Principal Investigator, Retinal Consultants of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E10030-003
Record Dates: First submitted 2014-03-27; First posted 2015-10-30 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — Ranibizumab; Bevacizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altering regimens of Fovista™and Anti-VEGF Therapy (Experimental): All subjects will be treated with Fovista™ 1.5 mg/eye in combination with anti-VEGF therapy.
  The following doses of Anti-VEGF therapy will be delivered based on the Investigator's discretion:
  * Lucentis® 0.5 mg/eye
  * Avastin® 1.25 mg/eye
  * Eylea® 2 mg/eye
  Subjects will be treated with Fovista™ and Anti-VEGF therapy every month for the first three months.
  The regimen for administration of each intravitreal agent will be as follows:
  Injection Day #1-Administration of Fovista™ 1.5mg/eye
  Injection Day #2-Administration of Fovista™ 1.5mg/eye followed by anti-VEGF therapy after Fovista™ injection
  The same regimen will be delivered monthly until the subject reaches maximum visual acuity benefit. Maximum visual acuity is defined as no increase in ETDRS visual acuity at two consecutive visits.
  Subsequent re-treatment with the Anti-VEGF therapy will use a PRN ("as-needed") regimen based on protocol specified retreatment criteria.
  Interventions: Drug: Fovista™; Drug: Lucentis®; Drug: Avastin®; Drug: Eylea®

INTERVENTIONS:
Drug: Fovista™ — Anti-PDGF-B pegylated aptamer
Drug: Lucentis® — Anti-VEGF
Drug: Avastin® — Anti-VEGF
Drug: Eylea® — Anti-VEGF

SUMMARY:
The objectives of this study are to establish the safety and tolerability of intravitreous administration of altering regimens of Fovista™ (Anti-PDGF-B pegylated aptamer) administered in combination with Anti-VEGF therapy (Lucentis®, Avastin® or Eylea®) in subjects with subfoveal neovascular age-related macular degeneration.

Subjects will be treated with Fovista™ and Anti-VEGF therapy every month for the first three months. Retreatment with Fovista™ and Anti-VEGF will occur if the following findings are present PER INVESTIGATOR DISCRETION:

* ≥ 5 ETDRS letters loss OR;
* Significant hemorrhage OR;
* New or increased RPE elevation consistent with increased disease activity OR;
* Increased neovascular lesion size OR;
* New or increased foveal intraretinal fluid

If anti-VEGF re-treatment is not administered based on the re-treatment criteria noted above, Fovista™ anti-PDGF therapy MUST be administered at a minimum of every 3 months (as monotherapy).

Therefore, subjects will be treated with Fovista™ or Anti-VEGF therapy for a total of 3-24 administrations.

ELIGIBILITY:
Inclusion Criteria:

* Active subfoveal choroidal neovascularization (CNV) due to AMD.
* Best corrected visual acuity in the study eye between 20/40 and 20/400, inclusive. The VA must be re-confirmed at Day 1 prior to randomization.
* Active CNV must compromise at least 25% of the lesion as measured on fluorescein angiogram (including blood, neovascularization, and scar/atrophy)
* Presence on OCT of subretinal hyper-reflective material (SHRM) within the central 1 mm subfield; SHRM is defined as hyper-reflective material located external to the outer retina and internal to the RPE, or, when the RPE is not well defined, internal to Bruch's membrane.
* Clear ocular media and adequate pupillary dilatation to allow collection of fundus photographs and fluorescein angiograms of a sufficient quality to
* Subjects of either gender aged ≥ 50 years.
* Women must agree to be using two forms of effective contraception, be post-menopausal for at least 12 months prior to trial entry, or surgically sterile; if of child-bearing potential, a serum pregnancy test must be performed within 14 days prior to the first injection with a negative result. The two forms of effective contraception must be implemented during the trial and for at least 60 days following the last dose of test medication.
* Provide written informed consent.
* Ability to comply with study and follow-up procedures and return for all trial visits.

Exclusion Criteria:

* More than 50% of the total lesion size made up of scarring or atrophy as determined by fundus photography with or without fluorescein angiography, with or without OCT. Subjects with any subfoveal scar or subfoveal atrophy directly below the center of the fovea are excluded.
* More than 50% of the total lesion size consisting of subretinal hemorrhage.
* Presence of retinal angiomatous proliferation (RAP).
* Presence of significant serous pigment epithelial detachments (PEDs), such as large PEDs that constitute greater than 50% of the total lesion or have a vertical height of ≥ 400 µm. Presence of pure PED without subretinal hyper-reflective material.
* Presence of pigment epithelial tears or rips.
* Presence of intraocular inflammation (≥ trace cell or flare), significant epiretinal membrane (causing distortion of macular anatomy and/or opacification), significant vitreomacular traction (causing distortion of macular anatomy), macular hole or vitreous hemorrhage.
* Aphakia or absence of the posterior capsule. Absence of an intact posterior capsule is allowed if it occurred as a result of YAG laser posterior capsulotomy in association with prior posterior chamber IOL implantation.
* History of idiopathic or autoimmune-associated uveitis in either eye.
* Significant media opacities, including cataract, which might interfere with visual acuity, assessment of toxicity, or fundus photography in the study eye. Subjects should not be entered if there is likelihood that they will require cataract surgery in the study eye in the next 12 months.
* Presence of other causes of choroidal neovascularization, including pathologic myopia (spherical equivalent of -8 diopters or more, or axial length of 25mm or more), the ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis.
* Any intraocular surgery or thermal laser within three (3) months of trial entry. Any prior thermal laser in the macular region, regardless of indication.
* Any ocular or periocular infection in the past twelve (12) weeks.
* History of any of the following conditions or procedures in the study eye: Rhegmatogenous retinal detachment, pars plana vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant.
* Previous therapeutic radiation in the region of the study eye. • History of other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
* History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV - see Appendix 17.5), history or clinical evidence of unstable angina, acute coronary syndrome, myocardial infarction or coronary artery revascularization within 6 months, or ventricular tachyarrythmias requiring ongoing treatment.
* Stroke (within 12 months of trial entry).
* Any major surgical procedure within one month of trial entry.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Safety endpoints include adverse events, vital signs, ophthalmic variables [ophthalmic examination, intraocular pressure (IOP), fluorescein angiogram (FA), optical coherence tomography (OCT)], ECG, and laboratory variables. | Month 24

SECONDARY OUTCOMES:
Mean change in amount of fibrosis as assessed by fundus photography and OCT evaluation. | Month 24

CONTACTS AND LOCATIONS:
Locations (1):
- Retinal Consultants of Arizona, Phoenix, Arizona, United States